CLINICAL TRIAL: NCT05452538
Title: Autotransfusion Versus Transfusion in Cancer Surgery
Acronym: ATTRACS
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ATTRACS
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hemorrhage; Cancer Surgery; Transfusion
Keywords: intraoperative blood salvage; cancer surgery; pharmacoeconomic analysis; transfusion
MeSH Terms: conditions — Hemorrhage | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer surgery: all adult patients operated at the Léon Bérard Centre for cancer surgery (excluding endoscopy, interventional radiology, brachytherapy, vascular access)
  Interventions: Device: Transfusion

INTERVENTIONS:
Device: Transfusion — Data from patients who were transfused at the Centre Léon Bérard from the day of surgery to the 10th postoperative day will be analyzed.

SUMMARY:
Acute bleeding is one of the most frequent intraoperative adverse events and is burdened with a significant morbidity and mortality rate.

The only available treatment for severe exsanguination is homologous transfusion, but this is itself complicated by side effects.

Nevertheless, systems exist allowing the recovery, treatment and intraoperative reinjection of lost blood, thus limiting transfusions.

DETAILED DESCRIPTION:
Acute bleeding is one of the most frequent intraoperative adverse events and is burdened with a significant morbidity and mortality rate.

The only available treatment for severe exsanguination is homologous transfusion, but this is itself complicated by side effects (immunosuppression, increased rate of carcinological recurrence...).

Nevertheless, systems exist allowing the recovery, treatment and intraoperative reinjection of lost blood, thus limiting transfusions.

The aim of this work is to collect and analyze the estimated bleeding and the hemoglobin level of patients who underwent an intermediate or major operation in the general block of the Centre Léon Bérard in 2021 and who were transfused within 10 days of this operation.

In the first stage of data analysis, the investigators will collect data related to perioperative transfusion currently performed at the Centre Léon Bérard (year 2021).

Then, a pharmacoeconomic analysis will be carried out with an evaluation of the cell salvage technique by mini-HTA (Health Technology Assessment) type (clinical benefit, patient safety, target population, robustness of clinical evidence, budgetary impact, amount of investment, impact in terms of human resources (training), efficiency) with the objective of helping the Centre Léon Bérard management to make a decision.

ELIGIBILITY:
Inclusion Criteria:

* Surgery at the Centre Léon Bérard in 2021
* transfusion from the day of surgery to the 10th postoperative day

Exclusion Criteria:

* Digestive endoscopy, interventional radiology, brachytherapy
* Vascular access only
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients who underwent surgery at the Centre Léon Bérard in 2021 and were transfused from the day of surgery to the 10th postoperative day
Sampling Method: Non-Probability Sample
Enrollment: 5808 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
number of annual uses of the intraoperative blood recovery system | Up to 1 year
  number of annual uses (at the Centre Léon Bérard in 2021) of the intraoperative blood recovery system in the indications validated by the French High Authority for Health

SECONDARY OUTCOMES:
annual cost for the Centre Léon Bérard of the transfusion strategy. | Up to 1 year
  Pharmacoeconomic analysis will be performed with an evaluation of the Cell-Saver mini-Health Technology Assessment technique (clinical benefit, patient safety, target population, robustness of clinical evidence, budgetary impact, investment amount, impact in terms of human resources (training), efficiency)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein AA, Bailey CR, Charlton AJ, Evans E, Guckian-Fisher M, McCrossan R, Nimmo AF, Payne S, Shreeve K, Smith J, Torella F. Association of Anaesthetists guidelines: cell salvage for peri-operative blood conservation 2018. Anaesthesia. 2018 Sep;73(9):1141-1150. doi: 10.1111/anae.14331. Epub 2018 Jul 10. PMID 29989144
- [Background] Waters JH, Yazer M, Chen YF, Kloke J. Blood salvage and cancer surgery: a meta-analysis of available studies. Transfusion. 2012 Oct;52(10):2167-73. doi: 10.1111/j.1537-2995.2011.03555.x. Epub 2012 Feb 10. PMID 22321196
- [Background] Ubee SS, Manikandan R, Gudimetla AR, Singh G. Cost benefits of intraoperative cell salvage in radical cystectomy. Indian J Urol. 2010 Apr;26(2):196-9. doi: 10.4103/0970-1591.65386. PMID 20877596
- [Background] Araujo RL, Pantanali CA, Haddad L, Rocha Filho JA, D'Albuquerque LA, Andraus W. Does autologous blood transfusion during liver transplantation for hepatocellular carcinoma increase risk of recurrence? World J Gastrointest Surg. 2016 Feb 27;8(2):161-8. doi: 10.4240/wjgs.v8.i2.161. PMID 26981190